CLINICAL TRIAL: NCT02020863
Title: Closed-Loop Fluid Administration System Using Hemodynamic Monitors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Maxime Cannesson, Professor, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCIANES03
Record Dates: First submitted 2013-12-19; First posted 2013-12-25 (Estimated); Results first posted 2016-05-27 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-04

CONDITIONS: Intraoperative Volume Status; Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Closed Loop (Experimental): Study patients will receive a baseline crystalloid infusion of 3 cc/kg/hr and all additional fluid management will be performed via a closed loop (automated) system that will determine rate, amount, and timing of fluid administration.
  Interventions: Device: Closed Loop

INTERVENTIONS:
Device: Closed Loop — Fluid management in the closed loop group will be performed via a closed loop (automated) system that will use an infusion pump (Q-Core) and a controller (a computer run index and algorithm developed by Sironis) to make frequent, regular and accurate adjustments to the amount of fluid the patient receives using feedback from standard operating room monitors.

SUMMARY:
The purpose of this study is to evaluate the feasibility of a closed-loop (automated) fluid administration system to deliver fluids using feedback from standard operating room hemodynamic monitors. In standard anesthesia care the rate of IV fluid administration to the patient is determined by the anesthesiologist caring for the patient. In this study protocol, the rate of fluid administration will be determined instead by the closed-loop (automated) control system under the supervision of the anesthesiologist. The system will independently decide when to give fluid and at what rate; the supervising anesthesiologist will monitor the system to ensure appropriate volumes are being delivered and to intervene if necessary.

DETAILED DESCRIPTION:
In our protocol we will test the hypothesis that closed-loop fluid administration can maintain higher cardiac stroke volume (shown to improve patient outcomes after surgery) than anesthesiologist management. We have shown this to be the case in multiple simulation studies and in-vivo animal studies, but not yet experimentally in a clinical setting. Investigators will recruit their patients from the surgical record that that require cardiac output monitoring undergoing surgery and require mechanical ventilation and consent to participate in the study will be included in the study. They will receive standard patient care in that in no way will their anesthetic or surgical procedure will be altered as part of the study, with the exception of fluid administration. Fluids are usually given to a patient based on the physician's discretion. As part of the study patients will receive fluid management via a closed loop (automated) system that will use an infusion pump (Q-Core) and a controller (a computer run index and algorithm developed by Sironis) to make frequent, regular and accurate adjustments to the amount of fluid the patient receives using feedback from standard operating room monitors at UCI). Data from this study will be retrospectively compared to subjects case matched to evaluate differences in cardiac output, total fluid given, and patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (over the age of 18)
* Subjects undergoing elective major, abdominal surgery
* Subjects requiring general anesthesia and mechanical ventilation
* Subjects requiring cardiac output monitoring and an arterial line

Exclusion Criteria:

* Subjects under 18 years of age
* Subjects not undergoing surgery
* Subjects not requiring general anesthesia or mechanical ventilation
* Subjects not requiring cardiac output monitoring or an arterial line
* Subjects who are pregnant
* Subjects without the capacity to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maxime Cannesson, MD, PhD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine Medical Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rinehart J, Liu N, Alexander B, Cannesson M. Review article: closed-loop systems in anesthesia: is there a potential for closed-loop fluid management and hemodynamic optimization? Anesth Analg. 2012 Jan;114(1):130-43. doi: 10.1213/ANE.0b013e318230e9e0. Epub 2011 Sep 29. PMID 21965362
- [Background] Bednarski P, Siclari F, Voigt A, Demertzis S, Lau G. Use of a computerized closed-loop sodium nitroprusside titration system for antihypertensive treatment after open heart surgery. Crit Care Med. 1990 Oct;18(10):1061-5. doi: 10.1097/00003246-199010000-00002. PMID 2209031
- [Background] Colvin JR, Kenny GN. Development and evaluation of a dual-pump microcomputer-based closed-loop arterial pressure control system. Int J Clin Monit Comput. 1989 Jan;6(1):31-5. doi: 10.1007/BF01723370. PMID 2723513
- [Background] Blankenship HB, Wallace FD, Pacifico AD. Clinical application of closed-loop postoperative autotransfusion. Med Prog Technol. 1990 May;16(1-2):89-93. PMID 2138701
- [Background] Bowman RJ, Westenskow DR. A microcomputer-based fluid infusion system for the resuscitation of burn patients. IEEE Trans Biomed Eng. 1981 Jun;28(6):475-9. doi: 10.1109/TBME.1981.324822. No abstract available. PMID 7287047
- [Background] Chaisson NF, Kirschner RA, Deyo DJ, Lopez JA, Prough DS, Kramer GC. Near-infrared spectroscopy-guided closed-loop resuscitation of hemorrhage. J Trauma. 2003 May;54(5 Suppl):S183-92. doi: 10.1097/01.TA.0000064508.11512.28. PMID 12768123
- [Background] DeBey RK, Westenskow DR, Jordan WS, McJames SW. A urine based control system for fluid infusion. Biomed Sci Instrum. 1987;23:195-8. No abstract available. PMID 3607171
- [Background] Rinehart J, Alexander B, Le Manach Y, Hofer C, Tavernier B, Kain ZN, Cannesson M. Evaluation of a novel closed-loop fluid-administration system based on dynamic predictors of fluid responsiveness: an in silico simulation study. Crit Care. 2011;15(6):R278. doi: 10.1186/cc10562. Epub 2011 Nov 23. PMID 22112587
- [Background] Rinehart J, Lee C, Cannesson M, Dumont G. Closed-loop fluid resuscitation: robustness against weight and cardiac contractility variations. Anesth Analg. 2013 Nov;117(5):1110-8. doi: 10.1213/ANE.0b013e3182930050. PMID 23835454
- [Background] Rinehart J, Lee C, Canales C, Kong A, Kain Z, Cannesson M. Closed-loop fluid administration compared to anesthesiologist management for hemodynamic optimization and resuscitation during surgery: an in vivo study. Anesth Analg. 2013 Nov;117(5):1119-29. doi: 10.1213/ANE.0b013e3182937d61. PMID 23835453
- [Background] Pearse R, Dawson D, Fawcett J, Rhodes A, Grounds RM, Bennett ED. Early goal-directed therapy after major surgery reduces complications and duration of hospital stay. A randomised, controlled trial [ISRCTN38797445]. Crit Care. 2005;9(6):R687-93. doi: 10.1186/cc3887. Epub 2005 Nov 8. PMID 16356219
- [Background] Forget P, Lois F, de Kock M. Goal-directed fluid management based on the pulse oximeter-derived pleth variability index reduces lactate levels and improves fluid management. Anesth Analg. 2010 Oct;111(4):910-4. doi: 10.1213/ANE.0b013e3181eb624f. Epub 2010 Aug 12. PMID 20705785
- [Background] Rinehart J, Chung E, Canales C, Cannesson M. Intraoperative stroke volume optimization using stroke volume, arterial pressure, and heart rate: closed-loop (learning intravenous resuscitator) versus anesthesiologists. J Cardiothorac Vasc Anesth. 2012 Oct;26(5):933-9. doi: 10.1053/j.jvca.2012.05.015. Epub 2012 Jul 12. PMID 22795172
- [Derived] Rinehart J, Lilot M, Lee C, Joosten A, Huynh T, Canales C, Imagawa D, Demirjian A, Cannesson M. Closed-loop assisted versus manual goal-directed fluid therapy during high-risk abdominal surgery: a case-control study with propensity matching. Crit Care. 2015 Mar 19;19(1):94. doi: 10.1186/s13054-015-0827-7. PMID 25888403
- [Derived] Joosten A, Huynh T, Suehiro K, Canales C, Cannesson M, Rinehart J. Goal-Directed fluid therapy with closed-loop assistance during moderate risk surgery using noninvasive cardiac output monitoring: A pilot study. Br J Anaesth. 2015 Jun;114(6):886-92. doi: 10.1093/bja/aev002. Epub 2015 Feb 17. PMID 25690834
- See also: Related info — http://www.sironis.com/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Closed Loop
Started | 40
Completed | 35
Not Completed | 5
Not completed — Discovery of Metastatic disease | 4
Not completed — Team chose not to place an a line | 1

BASELINE CHARACTERISTICS:
Arm/Group | Closed Loop
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 35
Specific Surgical procedure [Number; unit: participants]
  Whipple | 9
  Whipple + additional | 8
  Distal pancreatectomy | 5
  Liver resection | 10
  Complex cholecystectomy | 3
ASA Physical Status patient classification [Number; unit: participants] — ASA II A patient with mild systemic disease Mild diseases only without substantive functional limitations.
  ASA III A patient with severe systemic disease Substantive functional limitations; One or more moderate to severe diseases.
  ASA IV A patient with severe systemic disease that is a constant threat to life Examples include (but not limited to): recent ( < 3 months) MI, CVA, TIA, or CAD/stents, ongoing cardiac ischemia or severe valve dysfunction, severe reduction of ejection fraction, sepsis, DIC, ARD or ESRD not undergoing regularly scheduled dialysis
  participants
    2 | 1
    3 | 28
    4 | 6
Stroke Volume Index [Mean (Standard Deviation); unit: ml per meter-squared] | 44 (10)

OUTCOME MEASURES:

1. Primary Outcome: Fluid Status During Surgery
Description: The primary outcome between groups is preload independence, defined as % case time where Stroke Volume Variation (SVV) is ≤12%.
Time Frame: Duration of Surgery, up to 8 hours
Population: Closed Loop Study population at Stroke Volume Variation (SVV) ≤12%
Measure: Mean (Standard Deviation); unit: percentage of case time
Arm/Group | Closed Loop
Number analyzed (Participants) | 40
percentage of case time | 95 (6)

ADVERSE EVENTS:
Arm/Group | Closed Loop
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No